CLINICAL TRIAL: NCT00085280
Title: A Pilot Study to Determine if Downstream Markers of EGFR Linked Signaling Pathways Predict Response to OSI-774 (Erlotinib) in the First-Line Treatment of Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Erlotinib in Treating Patients With Stage IIIB, Stage IV, or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03147; NCI-2012-03147 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA021115 (NIH); CDR0000368459; ECOG-E3503; E3503 (Other: Eastern Cooperative Oncology Group); E3503 (Other: CTEP)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

ARMS (1):
- Treatment (erlotinib hydrochloride) (Experimental): Patients receive oral erlotinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Patients complete the Smoking Status Survey, a questionnaire regarding smoking habits, at baseline, and then every 3 months during study treatment.
  Interventions: Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial is studying how well erlotinib works in treating patients with stage IIIB, stage IV, or recurrent non-small cell lung cancer. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Prospectively identify downstream markers of EGFR linked signaling pathways that are predictive of response to OSI-774 (Erlotinib) in this population.

SECONDARY OBJECTIVES:

I. Estimate antitumor objective response rate per RECIST. II. Estimate disease control rate (CR+PR+SD). III. Estimate time to progression and overall survival. IV. Estimate if a grade 2 rash is a predictor of response to OSI-774 (Erlotinib) and of patient survival.

V. Assess safety profile of OSI-774 (Erlotinib) in this population. VI. To determine whether smoking status is linked to outcome for advanced NSCLC patients treated with OSI-774 (Erlotinib).

OUTLINE: This is a pilot, multicenter study.

Patients receive oral erlotinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients complete the Smoking Status Survey, a questionnaire regarding smoking habits, at baseline, and then every 3 months during study treatment.

After completion of study treatment, patients are followed every 3 months for 2 years, and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 129 patients will be accrued for this study within 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed NSCLC
* Patients must have diagnostic specimen available on paraffin-embedded block
* Patients must have advanced NSCLC (stage IIIB with a malignant pleural effusion or IV disease, or recurrent disease)
* Patients must not have received prior chemotherapy or targeted therapy for metastatic disease, including no prior EGFR inhibitor; patient may have received adjuvant chemotherapy for early stage disease (IB-IIIA), or chemo/XRT for stage IIIA or IIIB disease, provided s/he meets all of the following:

  * It has been at least 6 months since completion of patient's adjuvant chemotherapy for early stage disease (IB-IIIA) or chemo/XRT for stage IIIA or IIIB disease
  * Patient now has advanced disease
* Patients must have measurable disease per RECIST criteria; all sites of disease must be assessed within 4 weeks prior to registration
* Creatinine < 1.5 mg/dL or a creatinine clearance of > 50 mL/min
* SGOT(AST) and SGPT(ALT) < 2 x the institution's upper limit of normal
* Bilirubin < 1.5 mg/dL
* ANC > 1500/mm^3
* PLT > 100,000/mm^3
* Patients must have ECOG performance status 0, 1, or 2
* Patients with stable, treated brain metastases are eligible (defined as: patients with brain metastases must have been treated and are asymptomatic and are no longer taking corticosteroids)
* Patients with gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease, are ineligible
* Pregnant and breast feeding women are excluded from the study because the agent used in this study may be teratogenic to a fetus and there is no information on the excretion of the agents or their metabolites into breast milk
* Women of childbearing potential and sexually active males must agree to use an accepted and effective method of contraception (hormonal or barrier methods, abstinence) for the duration of the study
* HIV positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with OSI-774 (Erlotinib)
* Patients must not have had immuno, hormonal or radiation therapy within 2 weeks prior to entering the study; those who have not recovered from adverse events due to agents administered more than 2 weeks earlier are ineligible; previously irradiated areas can be considered "measurable disease" if there has been documented progression
* Patients must not have ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements
* Patients must not have serious non-healing wound, or bone fracture, or major surgical procedure within 21 days prior to study entry
* Patients taking Warfarin are eligible
* If the patient is taking Cyp3A4 inducers or inhibitors, they must be discontinued one week prior to starting OSI-774 (Erlotinib)
* Patients must not be enrolled in any other concurrent clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2004-09; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Response rates and distribution of the mitogen-activated protein kinase (MAPK)/extracellular-signal-regulated kinase (Erk)-phosphorylated expression groups based on the Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 5 years
  A Fisher's exact test with a two-sided 5% type I error rate will be calculated.

SECONDARY OUTCOMES:
Objective response rate based on the RECIST | Up to 5 years
Disease control rate (complete response [CR]+partial response [PR]+stable disease [SD]) | Up to 8 weeks
Time to progression | Date of entry on the study to the appearance of new metastatic lesions or objective tumor progression, up to 5 years
Overall survival | Up to 5 years
Toxicities associated with erlotinib hydrochloride, based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 | Up to 5 years
Relationship between clinical response and each of the markers using the semiquantitative histo-score method | Baseline
  Cox regression models will be used.
Effects of smoking status in terms of disease and survival | Up to 5 years
  Descriptive and summary statistics will be conducted on the smoking questionnaire data.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Brahmer, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Brahmer JR, Lee JW, Traynor AM, Hidalgo MM, Kolesar JM, Siegfried JM, Guaglianone PP, Patel JD, Keppen MD, Schiller JH. Dosing to rash: a phase II trial of the first-line erlotinib for patients with advanced non-small-cell lung cancer an Eastern Cooperative Oncology Group Study (E3503). Eur J Cancer. 2014 Jan;50(2):302-8. doi: 10.1016/j.ejca.2013.10.006. Epub 2013 Nov 15. PMID 24246704